CLINICAL TRIAL: NCT01407120
Title: Effects of NBP for Children of Divorce 15 Years Later
Brief Title: 15 Year Follow-up of New Beginnings Program for Divorced Families
Acronym: NBF15
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sharlene Wolchik/ Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01MH071707-04 (NIH); 5P30MH068685-05 (NIH)
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Mental Disorder; Substance Use
Keywords: Prevention; Divorce
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mother Program (Experimental): 11 session program focused on parenting skills
  Interventions: Behavioral: New Beginnings Program
- Mother Plus Child Program (Experimental): 11 session Mother Program focused on parenting skills plus 11 session Child program focused on child coping skills
  Interventions: Behavioral: New Beginnings Program
- Literature Control (No Intervention): Families received books on children's post-divorce adjustment

INTERVENTIONS:
Behavioral: New Beginnings Program — A preventive intervention for divorced families.
  Arms: Mother Plus Child Program; Mother Program

SUMMARY:
The project is a 15-year follow-up of 240 young adults whose families participated in an experimental evaluation of the New Beginnings Program (NBP), a preventive intervention for divorced families. The NBP was provided in late childhood; the follow-up occurred in young adulthood. Families were randomly assigned to one of three conditions: mother program (MP), dual-component mother and child program (MPCP), or literature-control (LC) condition. Programs were designed to change several putative mediators of children's post-divorce mental health problems using empirically-supported change strategies. The investigators expected that the NBP would have either main or risk by program interactive effects on mental health and substance use problems and disorders, developmental tasks, parent-young adult relationships, physical health problems, and competencies, such that YAs who participated in NBP will have better functioning than YAs in the control condition. The investigators expected that the NBP will have either main or risk by program interactive effects on mothers' mental health; those in the NBP are expected to have fewer mental health problems than those in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Divorced in past two years
* Female residential parent
* At least one 9-12 year-old child resided (at least 50%) with the mother
* Neither mother nor any child was currently in treatment for mental health problems
* Mother had not remarried nor planned to remarry during the program, and did not have a live-in boyfriend
* Custody was expected to remain stable
* Family resided within an hour drive of program site
* Mother and child could complete assessments in English
* Child was not learning disabled nor in special education
* If diagnosed with attention deficit disorder, child was taking medication

Exclusion Criteria:

* Child scored above 17 on the Children's Depression Inventory (CDI, endorsed an item indicating that s/he wanted to kill her/himself, or scored above the 97th percentile on the Externalizing Subscale (Child Behavior Checklist [CBCL])

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2006-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of mental health disorder | 15 year follow-up
  Incidence and number of internalizing, externalizing, and substance use disorders with onset of symptoms within the last nine years.

SECONDARY OUTCOMES:
Young Adult Substance Use | 15 year follow-up
  Frequency of substance use past month, and age of onset of regular drinking.
Internalizing and Externalizing Problems | 15 Year follow-up
  Number of internalizing and externalizing problems during the past 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene A Wolchik, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University: Prevention Research Center, Tempe, Arizona, United States

REFERENCES:
- [Background] Wolchik SA, Sandler IN, Millsap RE, Plummer BA, Greene SM, Anderson ER, Dawson-McClure SR, Hipke K, Haine RA. Six-year follow-up of preventive interventions for children of divorce: a randomized controlled trial. JAMA. 2002 Oct 16;288(15):1874-81. doi: 10.1001/jama.288.15.1874. PMID 12377086
- [Background] Wolchik SA, West SG, Sandler IN, Tein JY, Coatsworth D, Lengua L, Weiss L, Anderson ER, Greene SM, Griffin WA. An experimental evaluation of theory-based mother and mother-child programs for children of divorce. J Consult Clin Psychol. 2000 Oct;68(5):843-56. PMID 11068970
- [Derived] Elam KK, Sandler I, Wolchik S, Tein JY. Non-Residential Father-Child Involvement, Interparental Conflict and Mental Health of Children Following Divorce: A Person-Focused Approach. J Youth Adolesc. 2016 Mar;45(3):581-93. doi: 10.1007/s10964-015-0399-5. Epub 2015 Dec 21. PMID 26692236
- [Derived] Luecken LJ, Hagan MJ, Wolchik SA, Sandler IN, Tein JY. A Longitudinal Study of the Effects of Child-Reported Maternal Warmth on Cortisol Stress Response 15 Years After Parental Divorce. Psychosom Med. 2016 Feb-Mar;78(2):163-70. doi: 10.1097/PSY.0000000000000251. PMID 26465217
- [Derived] Herman PM, Mahrer NE, Wolchik SA, Porter MM, Jones S, Sandler IN. Cost-benefit analysis of a preventive intervention for divorced families: reduction in mental health and justice system service use costs 15 years later. Prev Sci. 2015 May;16(4):586-96. doi: 10.1007/s11121-014-0527-6. PMID 25382415
- [Derived] Luecken LJ, Hagan MJ, Mahrer NE, Wolchik SA, Sandler IN, Tein JY. Effects of a prevention program for divorced families on youth cortisol reactivity 15 years later. Psychol Health. 2015;30(7):751-69. doi: 10.1080/08870446.2014.983924. Epub 2014 Dec 3. PMID 25367835
- [Derived] Modecki KL, Hagan MJ, Sandler I, Wolchik SA. Latent profiles of nonresidential father engagement six years after divorce predict long-term offspring outcomes. J Clin Child Adolesc Psychol. 2015;44(1):123-36. doi: 10.1080/15374416.2013.865193. Epub 2014 Jan 31. PMID 24484456
- [Derived] Wolchik SA, Sandler IN, Tein JY, Mahrer NE, Millsap RE, Winslow E, Velez C, Porter MM, Luecken LJ, Reed A. Fifteen-year follow-up of a randomized trial of a preventive intervention for divorced families: effects on mental health and substance use outcomes in young adulthood. J Consult Clin Psychol. 2013 Aug;81(4):660-73. doi: 10.1037/a0033235. Epub 2013 Jun 10. PMID 23750466